CLINICAL TRIAL: NCT00006113
Title: A Phase II Trial of a MART-1/gp100/Tyrosinase Peptide-Pulsed Dendritic Cell Vaccine Treated With CD40 Ligand/Gamma Interferon With Subcutaneous IL-2 for Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy Followed by Biological Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068125 (10M-99-1); LAC-USC-10M991; NCI-G00-1837; NCI-T99-0102
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; aldesleukin; CD40 Ligand; Interferon-gamma; B-Cell Activating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: MART-1 antigen
Biological: aldesleukin
Biological: gp100 antigen
Biological: recombinant CD40-ligand
Biological: recombinant interferon gamma
Biological: recombinant interleukin-4
Biological: sargramostim
Biological: therapeutic autologous dendritic cells
Biological: therapeutic tumor infiltrating lymphocytes
Biological: tyrosinase peptide
Radiation: Candida albicans skin test reagent

SUMMARY:
RATIONALE: Vaccines made from melanoma cells may make the body build an immune response to kill tumor cells. Biological therapies such as interferon gamma and interleukin-2 use different ways to stimulate the immune system and stop cancer cells from growing. Combining vaccine therapy with biological therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying giving vaccine therapy together with interferon gamma and interleukin-2 in treating patients with stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical response rate and immune response in HLA-A2 positive patients with stage III or IV melanoma after receiving autologous dendritic cells pulsed with melanoma antigen peptides (MART-1:26-35, gp100:209-217, and tyrosinase:368-376) and treated ex vivo with CD40-ligand and interferon gamma, followed by interleukin-2 in vivo.
* Determine the toxicities of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients undergo leukapheresis to harvest autologous dendritic cells (ADCs). Melanoma peptides (MART-1:26-35, gp100:209-217, and tyrosinase:368-376) are pulsed separately onto ADCs, which are also treated ex vivo with CD40-ligand, interferon gamma, interleukin-4, sargramostim (GM-CSF), and Candida albicans skin test reagent. Patients receive each melanoma peptide pulsed ADC vaccine separately via 3 successive 10 minute infusions on day 1. Patients then receive interleukin-2 subcutaneously every 12 hours on days 2-6. Treatment repeats every 2 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks, then every 3 months for 2 years, then every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 21-41 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma

  * Measurable disease after attempted curative surgery
  * Unresectable stage III or IV uveal melanoma
  * Metastatic mucosal melanoma
* HLA-A2.1 positive
* No disease progression following high dose interleukin-2 (600,000 or 720,000 IU/kg every 8 hours)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 9.0 g/dL
* No coagulation disorders

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* Patients with documented or suspected coronary artery disease must undergo stress thallium test
* No major cardiovascular illness

Pulmonary:

* No major pulmonary illness

Immunologic:

* HIV negative
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative
* No history of uveitis or autoimmune inflammatory eye disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No major systemic infection
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior MART-1:26-35, gp100:209-217, or tyrosinase:368-376 antigens

Chemotherapy:

* At least 1 month since prior chemotherapy for melanoma

Endocrine therapy:

* No concurrent steroid therapy

Radiotherapy:

* At least 1 month since prior radiotherapy for melanoma

Surgery:

* See Disease Characteristics

Other:

* At least 1 month since prior adjuvant therapy for melanoma
* At least 1 month since other prior therapy for melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-06; Primary Completion 2003-05 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States